CLINICAL TRIAL: NCT01262079
Title: Evaluation of Influenza-Specific Immune Responses in Children and Adults During the 2010-2011 Influenza Season in the U.S.
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Vaccine Research Center, NIAID, NIH contact: Chief, Clinical Trials Core, Vaccine Research Center, NIAID, NIH
Other Study IDs: VRC 700; HHSN272201000049I (Other: Department of Health and Human Services)
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Influenza
Keywords: influenza; healthy volunteer; immunity; antibody; blood sample
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Plasma PBMC Whole-blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- Group 1: 6-15 years old
- Group 2: 16-25 years old
- Group 3: 26-35 years old
- Group 4: 36-45 years old
- Group 5: 46-55 years old
- Group 6: 56-65 years old
- Group 7: 66-75 years old
- Group 8: 76-85 years old
- Group 9: > 85 years old

SUMMARY:
This is a specimen collection protocol designed with the purpose of understanding the immune responses to influenza in children and adult subjects through collection of blood specimens and influenza medical history data. This protocol will allow the investigators to evaluate influenza-specific immune responses to a variety of influenza strains in a broad age range of the U.S. population early and late in the 2010-2011 influenza season. Immune responses will be evaluated using blood samples. The underlying hypothesis for this protocol is that the detailed characterization of immune responses to influenza in subjects from different age groups will further the understanding of immune responses cross-reactivity and advance development of influenza vaccines that are cross-reactive against old, new and re-emerging influenza strains.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 through 17 years and adults 18 years of age or older
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Able and willing to complete the informed consent/assent process
* Willing to donate blood for storage and for research, at least at three study visits
* Willing to have genetic tests performed on stored blood for research purposes

Exclusion Criteria:

* Known to be pregnant.
* Medical, psychiatric, occupational or other condition that, in the judgment of the site investigator, is a contraindication to protocol participation or impairs a subject's ability to give informed consent.
* Bleeding disorder diagnosis or any contraindications to blood drawing as assessed by the site investigator
* Immune system known to be compromised by HIV or other active infection, active cancer, or systemic immunosuppressive treatments.
* Seasonal influenza vaccine within the 12 weeks prior to enrollment.
* Another subject from the same household enrolled into the same age group.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy participants ages 6 years and older who are available for 3 clinic study visits over approximately eight months. Participants must be willing and able to donate blood for storage and research. Females must not be or become pregnant during the study. Multiple subjects from the same household may not be enrolled into the same age group.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Influenza-specific antibody responses | 2010-2011 influenza season
  To evaluate antibody responses to a panel of influenza strains across a broad age range of the U.S. population early as compared to late in the 2010-2011 influenza season.

SECONDARY OUTCOMES:
Influenza-specific T-cell responses | 2010-2011 influenza season
  To evaluate influenza-specific T-cell responses to a panel of influenza strains across a broad age range of the U.S. population early as compared to late in the 2010-2011 influenza season.

CONTACTS AND LOCATIONS:
Overall Officials: Barney S. Graham, M.D., Ph.D., Study Director — Chief: Clinical Trials Core
Locations (4):
- United States (4):
  - Hope Clinic of the Emory Vaccine Center, Decatur, Georgia
  - St. Louis University - Doisy Research Center, St Louis, Missouri
  - Cincinatti Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Wei CJ, Boyington JC, McTamney PM, Kong WP, Pearce MB, Xu L, Andersen H, Rao S, Tumpey TM, Yang ZY, Nabel GJ. Induction of broadly neutralizing H1N1 influenza antibodies by vaccination. Science. 2010 Aug 27;329(5995):1060-4. doi: 10.1126/science.1192517. Epub 2010 Jul 15. PMID 20647428
- [Background] Centers for Disease Control and Prevention (CDC). Serum cross-reactive antibody response to a novel influenza A (H1N1) virus after vaccination with seasonal influenza vaccine. MMWR Morb Mortal Wkly Rep. 2009 May 22;58(19):521-4. PMID 19478718
- See also: NIAID — http://www.niaid.nih.gov/Volunteer/VRC/Pages/default.aspx